CLINICAL TRIAL: NCT07114822
Title: Harnessing Online Peer Education For Fitness in People With Type II Diabetes
Brief Title: HOPE Intervention for Fitness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Sean D Young, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 7008
Record Dates: First submitted 2025-04-17; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOPE Group (Experimental): Group with Peer leaders
  Interventions: Behavioral: Harnessing Online Peer Education
- Control (No Intervention): Group without Peer Leaders

INTERVENTIONS:
Behavioral: Harnessing Online Peer Education — This group will have peer leaders that will engage participants in the groups. These peer leaders are those with type II diabetes that have over the recommended amount of exercise each week.
  Arms: HOPE Group

SUMMARY:
We will test the HOPE intervention on changing behavior of people to exercise more (take more steps each day).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Living in the US
* Self-report diagnosis of type II diabetes
* Has an app to track step count

Exclusion Criteria:

* On insulin or an injectable weight loss drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-21 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Step Count | 1 month
  Participants will take a screenshot of their monthly steps at baseline and after the 4-week intervention

SECONDARY OUTCOMES:
Average fasting glucose | 1 week
  Participants will be asked about their average fasting glucose in the past week at baseline and follow-up
HbA1c | Baseline
  Participants will self-report their most recent HbA1c
Change in weight and Body Mass Index (BMI) | 1 month
  Participants will self-report their weight and BMI measures

CONTACTS AND LOCATIONS:
Locations (1):
- UC Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No